CLINICAL TRIAL: NCT04885517
Title: Dynamic Transpulmonary Pressure in Covid-19 Pneumonia: Effects of Positive Pressure, Inspired Oxygen Fraction and Decubitus
Brief Title: Breathing Effort in Covid-19 Pneumonia: Effects of Positive Pressure, Inspired Oxygen Fraction and Decubitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Pietro Caironi, Professor, San Luigi Gonzaga Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2782
Record Dates: First submitted 2021-05-11; First posted 2021-05-13 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19 Pneumonia; Esophageal Pressure; Respiratory Drive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Spontaneous breathing, Venturi Mask FiO2 0.5, seated decubitus (Experimental): Patient will be evaluated after 20 minutes of spontaneous breathing, with FiO2 0.5 (Venturi Mask), during seated decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Spontaneous breathing, Non Rebreathing Mask, seated decubitus (Experimental): Patient will be evaluated after 20 minutes of spontaneous breathing, with FiO2 1 (Non Rebreathing Mask), during seated decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Continuous Positive Airway Pressure (CPAP) 7 cmH2O, FiO2 0.5, seated decubitus (Experimental): Patient will be evaluated after 20 minutes of CPAP (7 cmH2O), with FiO2 0.5, during seated decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Continuous Positive Airway Pressure (CPAP) 7 cmH2O, FiO2 0.5, supine decubitus (Experimental): Patient will be evaluated after 20 minutes of CPAP (7 cmH2O), with FiO2 0.5, during supine decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Continuous Positive Airway Pressure (CPAP) 7 cmH2O, FiO2 0.5, prone decubitus (Experimental): Patient will be evaluated after 20 minutes of CPAP (7 cmH2O), with FiO2 0.5, during prone decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Continuous Positive Airway Pressure (CPAP) 7 cmH2O, FiO2 1, seated decubitus (Experimental): Patient will be evaluated after 20 minutes of CPAP (7 cmH2O), with FiO2 1.0, during seated decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Continuous Positive Airway Pressure (CPAP) 12 cmH2O, FiO2 0.5, seated decubitus (Experimental): Patient will be evaluated after 20 minutes of CPAP (12 cmH2O), with FiO2 0.5, during seated decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter
- Continuous Positive Airway Pressure (CPAP) 12 cmH2O, FiO2 1, seated decubitus (Experimental): Patient will be evaluated after 20 minutes of CPAP (7 cmH2O), with FiO2 1.0, during seated decubitus. Respiratory, haemodynamics, and data on blood gas analysis will be obtained.
  Interventions: Device: Esophageal catheter

INTERVENTIONS:
Device: Esophageal catheter — Patients are equipped with an esophageal catheter: positioning is performed after accurate nasopharyngeal anesthesia with lidocaine

SUMMARY:
The study investigates the role of positive pressure, inspired oxygen fraction and different decubiti (seated, supine, prone) on breathing effort (as assessed by esophageal pressure swings) in Covid-19 pneumonia (at different disease stages) and in other causes of respiratory failure. The hypothesis is that positive pressure might be deleterious in terms of breathing effort if the main pathological mechanism associated with Sars-CoV-2 infection in the lung is not alveolar damage (as in other causes of respiratory failure) but vascular impairment as previously reported. The effects of high inspired oxygen fractions and decubiti might also be different with respect to other causes of respiratory failure.

DETAILED DESCRIPTION:
In spite of the overwhelming numbers of the current pandemic, many questions remain open regarding the pathophysiology of Covid-19 associated pneumonia. While some features of the disease (such as the oxygenation improvement associated with proning and/or continuous positive airway pressure) seem to line up with other causes of pneumonia characterized by primary alveolar damage, specific characteristics have been reported about Sars-CoV-2 lung infection which suggest a certain degree of parenchymal preservation and a predominant role of vascular impairment: the dissociation between lung volume and gas exchange, and the so called "happy hypoxemia" both evoke the possibility of mechanisms other than the loss of aeration as causes of hypoxia. Accordingly, evidence are now growing on the role of vascular dysregulation in this regard. It is probable, as previously put forward, that different stages exist in the disease which may account for the discordant findings of previous studies seeking to either associate or separate Covid-19 pneumonia and other causes of respiratory failure. In the present study we will compare the effects of three currently used approaches to improve gas exchange (continuous positive airway pressure, external oxygen administration and decubiti variations) in three different populations (1) early Covid-19 pneumonia, 2) severe late Covid-19 pneumonia and 3) non-Covid-19 pneumonia) in terms of breathing effort as assessed by esophageal pressure swings: our aim is to evaluate, in these populations, the real benefits (beyond the previously reported ones on gas exchange) of such strategies on lung rest. Our hypothesis is that, at least in the early stages of Covid-19 (and as opposed to other causes of respiratory failure), the application of positive pressure might be deleterious if no potential for recruitment, but rather a primary vascular impairment, is associated with hypoxia. If this will be the case the same (or a similar) degree of oxygenation improvement and a safer pattern of ventilation might be attained with the simple administration of oxygen or decubiti variations without the application of positive pressure, thus completely changing the current standards for the treatment of Covid-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Covid-19 early pneumonia)

* Age > 18
* Positive Sars-CoV 2 nasal swab
* interstitial pneumonia at either CT scan or chest X-ray
* Respiratory failure requiring CPAP for less than 48 hours
* FiO2 ≤0.5 and CPAP≤10 cmH2O

Group 2 (Covid-19 severe pneumonia)

* Age > 18
* Positive Sars-CoV 2 nasal swab
* interstitial pneumonia at either CT scan or chest X-ray
* Respiratory failure requiring CPAP
* Signs of severity with CPAP 10 cmH2O and FiO2 0.5: pulse oximetry (SpO2) ≤ 93% associated to either:

  * Dyspnea
  * Two or more signs of increased respiratory effort (respiratory rate ≥25 bpm, use of accessory inspiratory muscles , tirage, intercostal space depression, nasal flaring, expiratory abdominal efforts, PaCO2 < 35)

Group 3 (Non Covid-19 pneumonia)

* Age > 18
* Negative Sars-CoV 2 nasal swab
* CT scan or chest X-ray non compatible with Covid-19 associated pneumonia
* Respiratory failure requiring CPAP

Exclusion Criteria:

Group 1 (Covid-19 early pneumonia)

* Concomitant chronic pulmonary disease
* Chronic heart failure New York Heart Association (NYHA) 3-4
* Bacterial pulmonary associated infection (diagnosed or suspected)
* Pulmonary embolism
* Acute cardiogenic pulmonary edema
* Signs of severity with CPAP 10 cmH2O and FiO2 0.5: SpO2≤ 93% associated to either:

  * Dyspnea
  * Two or more signs of increased respiratory effort (respiratory rate ≥25 bpm, use of accessory inspiratory muscles , tirage, intercostal space depression, nasal flaring, expiratory abdominal efforts, PaCO2 < 35)
* At least one sign of respiratory fatigue/decompensation (pH<7.30 with PaCO2 >45, respiratory rate <15 bpm, paradoxal abdominal breathing, mental status alteration)

Group 2 (Covid-19 severe pneumonia)

* Concomitant chronic pulmonary disease
* Chronic heart failure NYHA 3-4
* Bacterial pulmonary associated infection (diagnosed or suspected)
* Pulmonary embolism
* Acute cardiogenic pulmonary edema
* At least one sign of respiratory fatigue/decompensation (pH<7.30 with PaCO2 >45, respiratory rate <15 bpm, paradoxal abdominal breathing, mental status alteration)

Group 3 (Non Covid-19 pneumonia)

* Concomitant chronic pulmonary disease
* Chronic heart failure NYHA 3-4
* Bacterial pulmonary associated infection (diagnosed or suspected)
* Pulmonary embolism
* Acute cardiogenic pulmonary edema
* At least one sign of respiratory fatigue/decompensation (pH<7.30 with PaCO2 >45, respiratory rate <15 bpm, paradoxal abdominal breathing, mental status alteration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressure swings at different levels of positive end-expiratory pressure (PEEP) | 160 minutes
  The main outcome of the study is represented by the difference in esophageal pressure swings (expiratory minus inspiratory) between the three levels of end expiratory pressure applied (0-7-12 cmH2O)

SECONDARY OUTCOMES:
Esophageal pressure swings at different levels of inspired oxygen fraction | 160 minutes
  One of the secondary outcomes of the study is represented by the difference in esophageal pressure swings (expiratory minus inspiratory) between the two levels of FiO2 applied (0.5-1)
Esophageal pressure swings at different decubiti | 160 minutes
  One of the secondary outcomes of the study is represented by the difference in esophageal pressure swings (expiratory minus inspiratory) between the three decubiti applied (seated, supine, prone)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Caironi, MD, Principal Investigator — San Luigi Gonzaga Hospital; Lorenzo Giosa, MD, Principal Investigator — San Luigi Gonzaga Hospital
Locations (1):
- A.O.U. San Luigi Gonzaga Di Orbassano, Orbassano, Italy/Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gattinoni L, Coppola S, Cressoni M, Busana M, Rossi S, Chiumello D. COVID-19 Does Not Lead to a "Typical" Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2020 May 15;201(10):1299-1300. doi: 10.1164/rccm.202003-0817LE. No abstract available. PMID 32228035
- [Result] Couzin-Frankel J. The mystery of the pandemic's 'happy hypoxia'. Science. 2020 May 1;368(6490):455-456. doi: 10.1126/science.368.6490.455. No abstract available. PMID 32355007
- [Result] Aliberti S, Radovanovic D, Billi F, Sotgiu G, Costanzo M, Pilocane T, Saderi L, Gramegna A, Rovellini A, Perotto L, Monzani V, Santus P, Blasi F. Helmet CPAP treatment in patients with COVID-19 pneumonia: a multicentre cohort study. Eur Respir J. 2020 Oct 15;56(4):2001935. doi: 10.1183/13993003.01935-2020. Print 2020 Oct. PMID 32747395
- [Result] Elharrar X, Trigui Y, Dols AM, Touchon F, Martinez S, Prud'homme E, Papazian L. Use of Prone Positioning in Nonintubated Patients With COVID-19 and Hypoxemic Acute Respiratory Failure. JAMA. 2020 Jun 9;323(22):2336-2338. doi: 10.1001/jama.2020.8255. PMID 32412581
- [Result] Chiumello D, Busana M, Coppola S, Romitti F, Formenti P, Bonifazi M, Pozzi T, Palumbo MM, Cressoni M, Herrmann P, Meissner K, Quintel M, Camporota L, Marini JJ, Gattinoni L. Physiological and quantitative CT-scan characterization of COVID-19 and typical ARDS: a matched cohort study. Intensive Care Med. 2020 Dec;46(12):2187-2196. doi: 10.1007/s00134-020-06281-2. Epub 2020 Oct 21. PMID 33089348
- [Result] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Result] Poston JT, Patel BK, Davis AM. Management of Critically Ill Adults With COVID-19. JAMA. 2020 May 12;323(18):1839-1841. doi: 10.1001/jama.2020.4914. No abstract available. PMID 32215647
- [Result] Gattinoni L, Giosa L, Bonifazi M, Pasticci I, Busana M, Macri M, Romitti F, Vassalli F, Quintel M. Targeting transpulmonary pressure to prevent ventilator-induced lung injury. Expert Rev Respir Med. 2019 Aug;13(8):737-746. doi: 10.1080/17476348.2019.1638767. Epub 2019 Jul 5. PMID 31274034
- [Result] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Result] Tonelli R, Fantini R, Tabbi L, Castaniere I, Pisani L, Pellegrino MR, Della Casa G, D'Amico R, Girardis M, Nava S, Clini EM, Marchioni A. Early Inspiratory Effort Assessment by Esophageal Manometry Predicts Noninvasive Ventilation Outcome in De Novo Respiratory Failure. A Pilot Study. Am J Respir Crit Care Med. 2020 Aug 15;202(4):558-567. doi: 10.1164/rccm.201912-2512OC. PMID 32325004
- [Result] Goligher EC, Jonkman AH, Dianti J, Vaporidi K, Beitler JR, Patel BK, Yoshida T, Jaber S, Dres M, Mauri T, Bellani G, Demoule A, Brochard L, Heunks L. Clinical strategies for implementing lung and diaphragm-protective ventilation: avoiding insufficient and excessive effort. Intensive Care Med. 2020 Dec;46(12):2314-2326. doi: 10.1007/s00134-020-06288-9. Epub 2020 Nov 2. PMID 33140181
- [Result] Apigo M, Schechtman J, Dhliwayo N, Al Tameemi M, Gazmuri RJ. Development of a work of breathing scale and monitoring need of intubation in COVID-19 pneumonia. Crit Care. 2020 Jul 31;24(1):477. doi: 10.1186/s13054-020-03176-y. No abstract available. PMID 32736637
- [Result] Vaporidi K, Akoumianaki E, Telias I, Goligher EC, Brochard L, Georgopoulos D. Respiratory Drive in Critically Ill Patients. Pathophysiology and Clinical Implications. Am J Respir Crit Care Med. 2020 Jan 1;201(1):20-32. doi: 10.1164/rccm.201903-0596SO. PMID 31437406
- [Result] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Derived] Giosa L, Collins PD, Sciolla M, Cerrone F, Di Blasi S, Macri MM, Davicco L, Laguzzi A, Gorgonzola F, Penso R, Steinberg I, Muraccini M, Perboni A, Russotto V, Camporota L, Bellani G, Caironi P. Effects of CPAP and FiO2 on respiratory effort and lung stress in early COVID-19 pneumonia: a randomized, crossover study. Ann Intensive Care. 2023 Oct 17;13(1):103. doi: 10.1186/s13613-023-01202-0. PMID 37847454